CLINICAL TRIAL: NCT06337474
Title: An Exploratory Clinical Study of the Safety and Efficacy of CD19 Chimeric Antigen Receptor NK Cell Injections for the Treatment of Refractory Primary Immune Thrombocytopenia
Brief Title: An Clinical Study of CD19 CAR NK Cells for the Treatment of Refractory Primary Immune Thrombocytopenia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changzhou No.2 People's Hospital (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Principal Investigator, Lu Xuzhang, Director, Department of Department of Hematology, Changzhou No.2 People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [2023]YLJSA089
Record Dates: First submitted 2024-03-19; First posted 2024-03-29 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Thrombocytopenia Alloimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 CAR NK cells (Experimental)
  Interventions: Drug: anti-CD19 CAR NK cells (KN5501)

INTERVENTIONS:
Drug: anti-CD19 CAR NK cells (KN5501) — Patients will receive Fludarabine (25 mg/m2 per day) and Cyclophosphamide (1000mg/m2 per day) on day -3. Doses of 9×10^9 cells, 13.5×10^9 anti-CD19 CAR NK cells (KN5501) will infused in each group using the dose-escalation strategy

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of CD19 CAR NK cells (KN5501) in patients with refractory immune thrombocytopenia. 9 patients are planned to be enrolled in the dose-escalation trial (9×10^9 cells, 13.5×10^9 cells). The primary objective of the study is to evaluation of the safety and feasibility of KN5501 for the treatment of relapsed/refractory B-cell related autoimmune diseases. The secondary objective is to evaluate evaluation of KN5501 for the treatment of refractory immune thrombocytopenia. The exploratory objective is to evaluate expansion, persistence and ability to deplete CD19 positive B cells of KN5501 in patients with refractory immune thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years old and ≤ 65 years old, male or female, subjects voluntarily participate in this clinical study and sign the Informed Consent Form (ICF);
2. Diagnosis of immune thrombocytopenia (UTP) (according to American Society of Hematology 2019 guidelines and International ITP Working Group);
3. Platelet count is decreased in routine blood tests at least two consecutive times, with no obvious abnormalities in the morphology of blood cells on microscopic examination of peripheral blood smears;
4. Spleen is not enlarged during screening;
5. The morphology of bone marrow cells in subjects is characterized by increased or normal megakaryocytes with impaired maturation;
6. Exclude other secondary thrombocytopenia: secondary thrombocytopenia due to autoimmune diseases, thyroid disorders, lymphoproliferative disorders, myelodysplastic syndromes (MDS), aplastic anemia (AA), various malignant blood disorders, neoplastic infiltrates, chronic liver disease, hypersplenism, common variable immunodeficiency disease (CVID), infections, vaccinations, etc.; thrombocytopenia; drug-induced thrombocytopenia; homozygous thrombocytopenia; thrombocytopenia during pregnancy; congenital thrombocytopenia and pseudothrombocytopenia. Thrombocytopenia due to consumption; drug-induced thrombocytopenia; isoimmune thrombocytopenia; thrombocytopenia in pregnancy; congenital thrombocytopenia and pseudothrombocytopenia;
7. Subjects with refractory ITP who are refractory to first-line therapeutic agents, thrombopoietic agents in second-line therapy, and rituximab, or who have had ineffective splenectomies/postoperative recurrences, and who undergo diagnostic reassessment and remain diagnosed with ITP;
8. Patients with refractory ITP: refractory to first-line therapeutic agents, thrombopoietic agents in second-line therapy, and rituximab; patients diagnosed with ITP despite unsuccessful splenectomy/postoperative recurrence on diagnostic reassessment
9. ECOG score ≤ 1;
10. Left ventricular ejection fraction (LVEF) ≥50% and no clinically significant pericardial effusion;
11. ≥ 4 weeks after subjects received last dose treatment (Radiotherapy, chemotherapy, monoclonal antibody therapy or other treatments);
12. NRT, antimalarial monotherapy, antimalarials in combination with OCS and/or immunosuppressants, combination of OCS and/or immunosuppressants.

Exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions;
2. Subjects with active infection receiving intravenous (IV) antibiotic treatment, or received intravenous (IV) antibiotic treatment within one week prior to anti-CD19 CAR NK Cell (KN5501) infusion;
3. Subjects with acquired and congenital immunodeficiency diseases;
4. Subjects with grade III or IV heart failure (NYHA classification);
5. History of epilepsy or other central nervous system (CNS) diseases;
6. History of severe herpes infections such as herpes encephalitis, ocular herpes, or diffuse herpes;
7. History of other primary malignant tumors except:

   a Cured non-melanoma skin cancer by surgical excision, for example basal cell carcinoma (BCC) ; b Cured primary malignant tumors, such as cervical cancer, superficial bladder cancer, breast cancer;
8. Signs of herpes or varicella zoster virus infection (specifically varicella, zoster) within 12 weeks prior to screening; history of any clinically significant cardiac, endocrine, hematologic, hepatic, immunologic, metabolic, urinary, pulmonary, neurologic, dermatologic, psychiatric, and renal disease or other significant medical condition, other than lupus, that prevents administration of BIIB059 (as determined by the investigator)
9. Females who are pregnant, lactating, or planning a pregnancy within six months;
10. History or current diagnosis of clinically significant non-ITP-induced thrombocytopenia
11. Subjects who have received other clinical trial treatment within 3 month;
12. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-08-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLTs) | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the Dose Limiting Toxicities (DLTs) of anti-CD19 CAR NK Cells for refractory immune thrombocytopenia
Treatment Emergent Adverse Events (TEAEs) | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the Treatment Emergent Adverse Events (TEAEs) of anti-CD19 CAR NK Cells for refractory immune thrombocytopenia

SECONDARY OUTCOMES:
Objective Response Rate of subjects | Time Frame: 2, 4, 8, 12, 16, 24, 28, 40 and 52 weeks after first infusion
  Objective Response is assessed according to definitions of International ITP Working Group. Objective Response Rate is defined as proportion of patients with PLT content.

CONTACTS AND LOCATIONS:
Locations (1):
- Changzhou Second People's Hospital, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No